CLINICAL TRIAL: NCT02898558
Title: Effect of Body Representation in Movement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Moss Rehabilitation Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 702940
Record Dates: First submitted 2016-09-08; First posted 2016-09-13 (Estimated); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Magnification hand size (Experimental): magnifying lenses used for 30 minutes daily for 14 days while completing a jigsaw puzzle
  Interventions: Behavioral: Magnification hand size; Device: magnifying lenses

INTERVENTIONS:
Behavioral: Magnification hand size — Participants will use magnifying lenses while completing a jigsaw puzzle for 30 min a day for 14 days.
Device: magnifying lenses

SUMMARY:
This study explores the possible implications of the increase in perceived body size for rehabilitation of motor functions. In a recent study we have tested if motor abilities of patients with stroke improve wearing magnifying lenses, showing that a beneficial effect of magnifying lenses can be observed in some patients. In the present study, we will identify 12 patients from this cohort who demonstrated an improvement greater than 10% in one or two motor task when wearing magnifying glasses. These participants will be invited to take part in a clinical study in which they will undergo a training phase: subjects will wear magnifying lenses at home for 30 minutes daily for 14 days while completing a jigsaw puzzle; a log will be kept to document participation. Participants' performance on different motor tasks will be assessed before, immediately after and 1 month after the training session. Standardized measures of motor performance will include the the Action Research Arm test and the Rivermead Assessment of Somatosensory Performance (RASP). In addition, participants will undergo grip strength, finger tapping tasks and a reaching and grasping task. We expect the repeated use of magnifying lenses to generate an improvement of patients' performance across tasks and this effect to be persistent in time.

DETAILED DESCRIPTION:
Altering the apparent size of a body part with magnifying changes tactile acuity, tactile distance judgments and pain perception.

In a recent study we have tested if motor abilities (grip strength, finger tapping and reaching and grasping) of patients with stroke improve wearing magnifying lenses. The results of this study showed that a beneficial effect of magnifying lenses on movement can be observed in some patients with stroke. The present study aims at following up these results and investigating the possible use of magnifying lenses in the rehabilitation to improve motor controls of stroke patients.

To pursuit this aim, we will identify 12 patients in our previous study cohort who demonstrated an improvement greater than 10% in the grip strength or finger tapping task when wearing magnifying glasses. These participants will be invited to take part in the present clinical study in which they will undergo a training phase: subjects will wear magnifying lenses at home for 30 minutes daily for 14 days while completing a jigsaw puzzle; a log will be kept to document participation. Participants' performance on different motor tasks will be assessed before, immediately after and 1 month after the training session. Standardized measures of motor performance will include the the Action Research Arm test and the Rivermead Assessment of Somatosensory Performance (RASP). In addition, participants will undergo grip strength (6 trials), finger tapping tasks (6 trials) and a reaching and grasping task, inn which they will be asked to reach and grasp 3 different objects (30 trials). We expect the repeated use of magnifying lenses to generate an improvement of patients' performance across task and this effect to be persistent in time.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from stroke who showed an improvement with magnifying lenses in our previous study.

Exclusion Criteria:

* Patients suffering from stroke who did not show an improvement with magnifying lenses in our previous study.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-09; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Action Research Arm test | Baseline, immediately after the training (two weeks) and after one month
  19 item measure of motor control (i.e. (grasp, grip, pinch, and gross arm movement). Max score is 57

SECONDARY OUTCOMES:
Rivermead Assessment of Somatosensory Performance | Baseline, immediately after the training (two weeks) and after one month
  Battery designed to test somatosensory functions, comprising of 7 subtests (sharp/dull discrimination, surface pressure touch, surface localization, sensory extinction, two-point discrimination, temperature discrimination, proprioception movement and direction discrimination). Max score for each subtest is 60, except for sensory extinction (max is 12) and two-point discrimination (fail or pass).
Grip strength | Baseline, immediately after the training (two weeks) and after one month
  A grip dynamometer measures participants' grip strength
Finger tapping | Baseline, immediately after the training (two weeks) and after one month
  Electronic tapping test measures participants' tapping rate of the index finger
Reach and grasping | Baseline, immediately after the training (two weeks) and after one month
  Motion tracking equipment used to measure participants kinematic parameters (movement time, peak velocity, grip aperture, etc.) when reaching and grasping 3 objects, for a total of 30 movements.

CONTACTS AND LOCATIONS:
Overall Officials: Branch Coslett, MD, Principal Investigator — University of Pennsylvania; Steven Jax, PhD, Study Director — MOSS S.p.A.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kennett S, Taylor-Clarke M, Haggard P. Noninformative vision improves the spatial resolution of touch in humans. Curr Biol. 2001 Aug 7;11(15):1188-91. doi: 10.1016/s0960-9822(01)00327-x. PMID 11516950
- [Background] Taylor-Clarke M, Jacobsen P, Haggard P. Keeping the world a constant size: object constancy in human touch. Nat Neurosci. 2004 Mar;7(3):219-20. doi: 10.1038/nn1199. Epub 2004 Feb 15. PMID 14966526
- [Background] Mancini F, Longo MR, Kammers MP, Haggard P. Visual distortion of body size modulates pain perception. Psychol Sci. 2011 Mar;22(3):325-30. doi: 10.1177/0956797611398496. Epub 2011 Feb 8. PMID 21303990
- [Background] Yozbatiran N, Der-Yeghiaian L, Cramer SC. A standardized approach to performing the action research arm test. Neurorehabil Neural Repair. 2008 Jan-Feb;22(1):78-90. doi: 10.1177/1545968307305353. Epub 2007 Aug 17. PMID 17704352
- [Background] Winward CE, Halligan PW, Wade DT. The Rivermead Assessment of Somatosensory Performance (RASP): standardization and reliability data. Clin Rehabil. 2002 Aug;16(5):523-33. doi: 10.1191/0269215502cr522oa. PMID 12194623